CLINICAL TRIAL: NCT03625856
Title: The Effect of Chlorella Vulgaris Supplementation on Glycemic Control, Lipid Profile and Anthropometric Measurements on Patients With Type 2 Diabetes Mellitus
Brief Title: The Effect of Chlorella Supplementation on Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behnood Abbasi (Other)
Responsible Party: Sponsor-Investigator, Dr. Behnood Abbasi, Clinical Professor, Islamic Azad University, Sanandaj
Organization: Islamic Azad University, Sanandaj (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.TUMS.EMRI.REC.1396.00195
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated into two groups; Chlorella and placebo groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is a double-blind, randomized controlled trial. Subjects will be randomly allocated into two groups and each one will receive the supplement (Chlorella Vulgaris) or placebo for 8 weeks. To prevent selection bias, the study participants, investigators and the laboratory staff will be all blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 1500 mg Chlorella Vulgaris capsule
  Interventions: Dietary Supplement: Chlorella Vulgaris
- Control (Placebo Comparator): 1500 mg placebo (starch)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Chlorella Vulgaris — Chlorella capsules 1500 mg/day
  Other Names: Algomed
  Arms: Intervention
Dietary Supplement: Placebo — Starch 1500 mg
  Arms: Control

SUMMARY:
Diabetes is a chronic disease and the prevalence of diabetes mellitus is rapidly increasing as a result of population ageing, urbanization and associated lifestyle changes. Recently, the use of natural products in chronic diseases such as diabetes has gained more attention. Chlorella is a single-celled green algae that contains essential nutrients including amino acids and fatty acids as well as some vitamins and minerals. There have been some studies on the effects of chlorella supplementation in chronic diseases such as NAFLD, prediabetes and diabetic mice, but none of them examined the effects of chlorella in patients with type 2 diabetes. Thus the present study designed to evaluate the effects of chlorella supplementation on glycemic control, lipid profile and anthropometric measurements in type 2 diabetic patients.

DETAILED DESCRIPTION:
This study is a double-blind, randomized controlled trial. 84 patients with type 2 diabetes are recruited. After informing the patients about this study and filling the consent letters, they are randomly assigned into intervention group (n=42) or placebo group (n=42) receiving 1500 mg chlorella Vulgaris or placebo daily for 8 weeks. Patients are asked not to change their regular physical activity, diet, medicine and dosage during the study. Anthropometric and blood pressure measurements are collected and 24-hour food intake recall, IPAQ physical activity, Pittsburgh Sleep Quality Assessment (PSQI) and Beck anxiety and depression questionnaires are filled by each patients at the beginning and end of the study. In addition, blood samples are collected at the beginning and end of the study to determine the changes of FBS, HbA1c, insulin concentration and insulin resistance (HOMA-IR) and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Tendency to participate
* Clinical diagnosis of T2DM
* Having T2DM for at least 1 year
* Range of HbA1c between 6.5% and 8.5%
* Triglyceride range lower than 300 mg/dl

Exclusion Criteria:

* Insulin dependent patients
* Smoking and alcohol consumption
* Patients with cardiovascular disease, liver disease, renal and thyroid diseases
* Pregnancy, lactation and menopause
* Intake of multivitamin and mineral supplements

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
HbA1c changes | Baseline and after 8 weeks
  Serum HbA1c concentration

SECONDARY OUTCOMES:
FBS changes | Baseline and after 8 weeks
  Serum glucose concentration
Insulin sensitivity changes | Baseline and after 8 weeks
  HOMA-IR
Triglyceride changes | Baseline and after 8 weeks
  Serum TG concentration
Total cholesterol changes | Baseline and after 8 weeks
  Serum TC concentration
HDL-Cholesterol changes | Baseline and after 8 weeks
  Serum HDL concentration
Weight change | Baseline and after 8 weeks
  Body weight of participants
Systolic blood pressure changes | Baseline and after 8 weeks
  Systolic blood pressure
Diastolic blood pressure changes | Baseline and after 8 weeks
  Diastolic blood pressure
Anxiety score changes | Baseline and after 8 weeks
  The beck anxiety inventory (BAI) is used for the evaluations. The total range of this 21 item questionnaire is from zero to 63. Responses are rated on a 4-point Likert scale and range from 0 (not at all) to 3 (severely). These points are summed and the total score of 0-7 for sub-scales is considered nonexistence or the least form of anxiety,8-15 slight,16-25 moderate and 26-63 indicate the severe form of it.
Depression score changes | Baseline and after 8 weeks
  The beck depression inventory (BDI) is used for the evaluations. The total range of this 21 item questionnaire is from zero to 40. BDI items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. These points are summed and the total score of 0-10 for sub-scales is considered normal,11-16 Mild mood disturbance,17-20 borderline clinical depression, 21-30 moderate depression, 31-40 severe depression and over 40 is considered extreme depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keshavarz, Ph.D., Principal Investigator — Islamic Azad University,Science and Research Branch
Locations (1):
- Amir Mahdi Hosseini, Tehran, Iran